CLINICAL TRIAL: NCT04149028
Title: Platelet Rich Plasma Injection Into Ovary of Patients With Premature Ovarian Insufficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman S Dawood, MD, Lecturer of Obstetrics and gynecology, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POFPRP
Record Dates: First submitted 2019-10-30; First posted 2019-11-04 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Premature Ovarian Failure
Keywords: Premature ovarian insuffiency; Infertility; PRP
MeSH Terms: conditions — Primary Ovarian Insufficiency; Infertility

STUDY DESIGN:
Intervention Model Description: All eligible patient will recieve the treatment with PRP
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRP injection (Experimental): injection of PRP inside ovary by the assistance of laparoscopy
  Interventions: Procedure: PRP injection inside the ovary by laparoscoy. The injection volume is 2 ml

INTERVENTIONS:
Procedure: PRP injection inside the ovary by laparoscoy. The injection volume is 2 ml — intraovarian injection of 2 mml of PRP by laparoscopic guide

SUMMARY:
All encountered cases with POI will be assessed and examined then investigated. Eligible cases will be included in the study

DETAILED DESCRIPTION:
Patients will be subjected to injection of autologous PRP inside the ovary about 0.5-1 mml by laparoscopy

ELIGIBILITY:
Inclusion Criteria:

* Premature ovarian insufficiency diagnosed by:
* FSH> 40 Amenorrhea Menopuasal symptoms Infertility

Exclusion Criteria:

* Refusal to participate Secondary POI due chemotherapy, surgery, or radiotherapy Previous treatment with PRP

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Resumption of ovarian hormonal function | 3-6 months
  Measurement of Estradiol level on Day 3 of cycle
Resumption of ovarian folliclugenesis | 3-6 months
  Assessment of the presence of oocytes by trans vaginal ultrasound on day 3

SECONDARY OUTCOMES:
Resumption of menstruation | 3-6 months
  Occurrence of Menstruation after secondary amenrorrhea by questionnaire
Fertility potential | 3-6 months
  Potential to get pregnant after ICSI procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Adel Elgergawy, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
we will decide later